CLINICAL TRIAL: NCT05734989
Title: Improving Screening and Therapy Provision Among Hispanics/Latinx at Risk for Chronic Kidney Disease
Brief Title: Improving Screening and Therapy for Hispanic/Latinx at Risk for CKD
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00112455
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes; Chronic Kidney Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hispanic/Latinx patients at risk for CKD: Adult patients in the Hispanic/Latinx Durham community screened for CKD
  Interventions: Diagnostic Test: BP; Diagnostic Test: HbA1c
- PCPs caring for Hispanic Latinx patients screened for CKD in the Durham Community: Primary Care Providers (PCPs) caring for Hispanic Latinx patients who agree to use the study guidelines and interventions for screening and monitoring their patients for CKD.
  Interventions: Behavioral: PCP Guidelines for Screening and Monitoring Hispanic/Latinx patients for CKD

INTERVENTIONS:
Diagnostic Test: BP — Blood pressure measurements and HbA1c tests will be conducted to identify participants with or at risk for high blood pressure and/or Type 2 Diabetes. Those identified will be referred to PCP for follow up/treatment.
  Groups: Hispanic/Latinx patients at risk for CKD
Diagnostic Test: HbA1c — HbA1c will screen to identify patients with Type 2 diabetes
  Groups: Hispanic/Latinx patients at risk for CKD
Behavioral: PCP Guidelines for Screening and Monitoring Hispanic/Latinx patients for CKD — Guidelines will be developed and provided to PCPs to use with their Hispanic/Latinx patients with or at risk for CKD.
  Groups: PCPs caring for Hispanic Latinx patients screened for CKD in the Durham Community

SUMMARY:
In this study, the investigators will utilize community organizations to screen Hispanics/Latino(a)s for kidney disease, diabetes, and other risk factors, and refer them for care with a PCP. Additionally, the investigators will implement an intervention in local health clinics to assist PCPs with screening and treating patients with diabetes.

Completion of the project will hopefully slow progression of kidney disease among Hispanic/Latino(a) patients in Durham, and the information gained will allow the investigators to eventually perform the intervention on a larger scale.

DETAILED DESCRIPTION:
The goals of this study are to (1) Increase rates of screening and monitoring of CKD and CKD risk factors for Hispanic/Latinx community members in Durham by utilizing existing community resources and screening events and (2) Pilot test a PCP-facing intervention to promote guideline concordant testing and evidence-based therapy provision for Hispanics/Latinx with T2D at community health centers, utilizing clinical champions and pharmacists. The investigators anticipate the study will identify patients with CKD or CKD risk factors and establish feasibility of the pilot intervention, which the investigators plan to ultimately apply on a large scale to reduce inequities and improve clinical outcomes among Hispanics/Latinx.

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

* Age 18 or older at time of screening
* Self-identifying as Hispanic/Latinx ethnicity.

Exclusion Criteria:

* Unable to be reached by telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aim 1:
  Adults in the Durham, NC Hispanic/Latinx community at risk for hypertension and/or CKD
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Number of patients referred to PCPs (Primary Care Providers) for CKD screening | 3 months from referral
  Increase rates of screening and monitoring of Chronic Kidney Disease (CKD) and CKD risk factors for Hispanic/Latinx community members in Durham by utilizing existing community resources and screening events

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sinclair, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/89/NCT05734989/ICF_000.pdf